CLINICAL TRIAL: NCT01325129
Title: Elastic Stable Intramedullary Nailing of Dislocated Clavicle Fractures in Children and Adolescents: Lessons Learned From the First 20 Patients
Brief Title: Elastic Stable Intramedullary Nailing of Dislocated Clavicle Fractures in Children
Acronym: ESIN clavicle
Status: Completed | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Martin M Kaiser, Consultant, University of Luebeck
Other Study IDs: DE814167313
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Dislocated Clavicular Fracture Treated With Elastic Stable Intramedullary Nailing
Keywords: ESIN; Clavicular Fracture; Dislocation; Children; Adolescents
MeSH Terms: conditions — Joint Dislocations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Most Clavicular Fractures in Children can be Treated Conservatively. Our Own Study showed a Benefit towards Much Lower Pain and Better Cosmesis in Adolescents when Treated with Elastic Stable Intramedullary Nailing.

The First 20 Patients Treated with this Method will be examined for Functional (CONSTANT and MURLEY-Score) and Cosmetic Results as well as Ultrasound-Morphology of both clavicles and Patients'satisfaction (CSS-8). Further on, all complications and problems will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Only Dislocated Shaft Fractures or Pseudarthrosis after Conservative Treatment of Dislocated CSF in Children and Adolescents Treated with Elastic Stable Intramedullary Nailing

Exclusion Criteria:

* Age > 17 years
* Pathologic fractures
* Lateral or Medial Fractures of the Clavicle

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Last 24 Patients we Treated with ESIN
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric Surgery University Hospital, Lübeck, Germany

REFERENCES:
- [Background] Prinz KS, Rapp M, Kraus R, Wessel LM, Kaiser MM. [Dislocated midclavicular fractures in children and adolescents: who benefits from operative treatment?]. Z Orthop Unfall. 2010 Jan;148(1):60-5. doi: 10.1055/s-0029-1186155. Epub 2009 Oct 19. German. PMID 20135591
- [Result] Rapp M, Prinz K, Kaiser MM. Elastic stable intramedullary nailing for displaced pediatric clavicle midshaft fractures: a prospective study of the results and patient satisfaction in 24 children and adolescents aged 10 to 15 years. J Pediatr Orthop. 2013 Sep;33(6):608-13. doi: 10.1097/BPO.0b013e31829d1a76. PMID 23812152